CLINICAL TRIAL: NCT06457334
Title: Effect of Helicobacter Pylori Eradication on Gastroesophageal RefIux Disease (GERD)
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Fergany Abdelhamid Elgamal, resident doctor, Assiut University
Other Study IDs: H.pylori eradication on GERD
Record Dates: First submitted 2024-05-27; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: GERD
Keywords: Helicobacter pylori
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Evaluate the effect of H.pylori eradication on Gastroesophageal-reflux disease and symptoms improvement

DETAILED DESCRIPTION:
HeIicobacter PyIori (H.pyIori) is a gram-negative spiral shaped bacterium that affects up to 50% of the population worldwide, with a higher prevalences in the developing countries,Gastroesophageal reflux disease (GERD) is a chronic gastrointestinal disorder characterized by the regurgitation of gastric contents into the esophagus, resulting in a significant economic burden in direct and indirect costs and adversely affects the quality of life.GERD is caused by multiple different mechanisms that can be intrinsic, structural, or both, leading to the disruption of the esophago-gastric junction barrier resulting in exposure of the esophagus to acidic gastric contents, Clinically, GERD typically manifests with symptoms of heartburn and regurgitation. It can also present in an atypical fashion with extra-esophageal symptoms such as chest pain, dental erosions, chronic cough, laryngitis, or asthma.The relationship between H. pylori and gastroesophageal reflux disease (GERD) is still unclear, and the effect of H. pylori eradication on GERD treatment is unknown.Several studies have shown the inverse relationship between the occurrence of GERD and H.pyIori infection, in particular an increased severity of the disease is documented in patients with pre-existing symptoms .It has been showed that a markedly resolution of dyspepsia in patients at whom the eradication therapy was successful when compared with subjects with a persistent infection

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed as GERD clinically and endscopically.

Exclusion Criteria:

* NO exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients diagnosed as GERD clinically and endscopically.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Eradication of Helicobacter pylori after triple therapy | 1\2024 to 12\2024
  H.pylori eradication will be assessed using the endoscope
Effect of Helicobacter pylori eradication on Gastroesophageal RefIux disease (GERD) syptomes | 1\2024 to 12\2024
  Evaluate the effect of H.pylori eradication on Gastroesophageal-reflux disease and correlate with GERD symptoms improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Saad Z Mahmoud, Professor, Study Director — Assiut University
Locations (1):
- Alrajhi Hospital, Asyut, Egypt

REFERENCES:
- [Background] Ceylan A, Kirimi E, Tuncer O, Turkdogan K, Ariyuca S, Ceylan N. Prevalence of Helicobacter pylori in children and their family members in a district in Turkey. J Health Popul Nutr. 2007 Dec;25(4):422-7. PMID 18402185